CLINICAL TRIAL: NCT05689918
Title: Gastroesophageal Reflux Symptoms and Help-seeking Behavior, Medication Use and Esophageal Cancer Awareness: Dutch Population-based Survey
Brief Title: Gastroesophageal Reflux Disease in the Dutch Population
Acronym: REFLUX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13720
Record Dates: First submitted 2022-11-30; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-11

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Rationale: Screening for esophageal adenocarcinoma (EAC) precursors and treating them may help to decrease mortality of this malignancy. To understand the size of the target population for potential EAC screening, insight in the prevalence of registered and unregistered individuals with gastro-esophageal reflux disease (GERD) symptoms is needed. Insight in public awareness of EAC will provide additional useful information for public communication strategies.

Objective: The aims of this study are to assess the prevalence of GERD symptoms and related help-seeking behavior, registered and unregistered medication use and awareness of esophageal cancer in the general Dutch population.

Study design: Cross-sectional population-based survey.

Study population: Dutch citizens aged 18-75 years.

Methods: Eligible individuals will be selected from the Dutch population registry (BRP) using simple random sampling. Invitations will be sent by postal mail with participants being directed to a digital survey.

Main study parameters/endpoints: The outcome variables are presence of current GERD symptoms, number of GERD patients that consulted a doctor, number of GERD patients using prescribed and/or over the counter (OTC) antacids, histamine-receptor antagonists (H2RAs) and proton pump inhibitors (PPIs), and awareness and beliefs about esophageal cancer. The association between socio-demographic background and outcome variables will also be evaluated.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will not directly benefit from participating in this study.

Nonetheless, participating in this study is not associated with any healthcare risks and the burden for the subjects is very low. The survey has a low burdensome nature and will take approximately 20 minutes to complete. All data will be pseudonymized, refusal to fill out the survey or desire to withdraw from the study will not have any consequences for the invited subject.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years

Exclusion Criteria:

* Unable to provide informed consent for any reason;
* Unable to fill out the digital survey for any reason.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dutch population registry, 'Basisregistratie Personen' (BRP).
Sampling Method: Probability Sample
Enrollment: 4719 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-03-07 (Estimated); Study Completion 2023-05-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of GERD symptoms (heartburn, regurgitation and/or dyspepsia) | 7 days
  The Dutch translation of the validated Reflux Disease Questionnaire will be used to measure this outcome.
Level of awareness of esophageal cancer risk factors and alarm symptoms | Baseline
  The awareness and beliefs about cancer (ABC) measure was adapted for this outcome. The alarm symptom module measures whether participants think dysphagia, change in stool pattern, change in appearance of a mole, weightloss and palpable lesions are alarm symptoms of cancer (yes/no/don't know). The risk factor module measures whether participants think alcohol, smoking, obesity, male sex, GERD symptoms, age>50y, familial esophageal cancer, hot drinks and radiation are risk factors for esophageal cancer on a 4 point scale (strongly disagree - strongly agree).

SECONDARY OUTCOMES:
Number of individuals that sought help for GERD (general practitioner/referral) | 20 years
  Participants with GERD will be asked whether they discussed their symptoms with their GP, whether they have been referred to a gastroenterologist or internist and what their reasons were for seeking help or not seeking help (answer options were based on qualitative research).
Number of individuals with GERD that used antacids, H2RAs and PPI's (prescribed) | 6 months
  Participants will be asked to indicate whether they used prescribed Omeprazol, Pantoprazol, Esomeprazol, Lansoprazol, Rabeprazol, Cimetidine, Famotidine, Nizatidine, Ranitidine, Sucralfate, Misoprostol, Antagel, Gastilox, Maalox, Gaviscon, Regla-pH, Rennie, Magnesiumhydroxide, Iberogast or A. Vogel Boldocynara in the past 6 months.
Number of individuals with GERD that used antacids, H2RAs and PPI's (over-the-counter) | 6 months
  Participants will be asked to indicate whether they used over-the-counter Omeprazol, Pantoprazol, Esomeprazol, Lansoprazol, Rabeprazol, Cimetidine, Famotidine, Nizatidine, Ranitidine, Sucralfate, Misoprostol, Antagel, Gastilox, Maalox, Gaviscon, Regla-pH, Rennie, Magnesiumhydroxide, Iberogast or A. Vogel Boldocynara in the past 6 months.
Beliefs about esophageal cancer | Baseline
  The awareness and beliefs about cancer (ABC) measure was adapted for this outcome. The beliefs module measures whether participants think esophageal cancer can be treated, can be cured, is a death sentence, can benefit from early detection and whether they would wish to know about de diagnosis on a 4 point Likerts scale (strongly disagree - strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Huibertse LJ, Sijben J, Peters Y, Siersema PD. Self-management and help-seeking behavior for gastroesophageal reflux symptoms: A population-based survey. World J Gastroenterol. 2026 Jan 14;32(2):112395. doi: 10.3748/wjg.v32.i2.112395. PMID 41551831